CLINICAL TRIAL: NCT00639431
Title: Study to Assess the Efficacy of Direct Observation and Mental Visualization of Foot Movements to Treat Bilateral Lower Limb Phantom Limb Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jack Tsao, MD, Neurologist, Walter Reed Army Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DCI P07-71044
Record Dates: First submitted 2007-12-04; First posted 2008-03-20 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Phantom Limb Pain
Keywords: phantom limb pain; limb amputation; Amputation; Phantom Limb; Pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Direct observation of a sequence of right foot movements performed by the experimenter while visualizing moving the amputated or phantom right foot.
  Interventions: Behavioral: direct observation
- 2 (Experimental): Direct observation of a sequence of left foot movements performed by the experimenter while visualizing moving the amputated or phantom left foot.
  Interventions: Behavioral: direct observation
- 3 (Experimental): Direct observation of a sequence of left and right foot movements performed by the experimenter while visualizing moving the amputated or phantom left and right feet.
  Interventions: Behavioral: direct observation
- 4 (Experimental): Mental visualization with closed eyes of a sequence movements performed with the right amputated or phantom foot.
  Interventions: Behavioral: mental visualization
- 5 (Experimental): Mental visualization with closed eyes of a sequence movements performed with the left amputated or phantom foot.
  Interventions: Behavioral: mental visualization
- 6 (Experimental): Mental visualization with closed eyes of a sequence movements performed with the left and right amputated or phantom feet.
  Interventions: Behavioral: mental visualization

INTERVENTIONS:
Behavioral: direct observation — direct observation of another person's foot moving
  Arms: 1; 2; 3
Behavioral: mental visualization — mentally imagining moving one's phantom foot/feet
  Arms: 4; 5; 6

SUMMARY:
Because bilateral lower extremity amputees do not have an intact limb for use with the mirror, we are now proposing to conduct a pilot trial of two treatments for phantom limb pain (PLP) - direct observation of another person's foot moving versus mental visualization. The trial will last for 4 months and during the first month data will be gathered daily on the number of episodes of phantom limb pain, the average length of episodes, and the average intensity of pain in each phantom leg. In addition, the rapidity of pain relief, the length of therapy needed to sustain long-lasting pain relief, and whether use of these two treatment methods during rehabilitation can provide sustained and/or permanent pain relief will be determined. This study will test the hypothesis that direct observation of a limb while performing phantom limb movements will reduce phantom limb pain more than mental visualization of the phantom limb alone in subjects who have sustained a traumatic bilateral lower limb amputation.

DETAILED DESCRIPTION:
A total of forty-two (42) subjects with bilateral lower extremity amputations will be enrolled. Subjects will be randomized for assignment into two treatment conditions: twenty-one (21) subjects will use direct observation of another person's foot movements while twenty-one (21) will use mental visualization of foot movements (which will serve as the control group). Subjects in each group will be further be randomized for assignment into six treatment groups: direct observation or mental visualization of right lower extremity movements alone, direct observation or mental visualization of left lower extremity movements alone, or direct observation or mental visualization of simultaneous bilateral lower extremity movements. Subjects will use their assigned therapy for 20 minutes daily. The subjects for this study will be recruited from the Walter Reed Army Medical Center (WRAMC) Amputee clinic. Up to sixty (50) subjects will be recruited and screened according to the inclusion and exclusion criteria since we expect that some may not qualify or drop-out sooner than the scheduled 4-month completion time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 70 years of age, active duty military, beneficiary, or retiree.
* Written informed consent and written authorization for use or release of health and research study information.
* Traumatic bilateral lower limb amputation.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Normal neurological examination.
* Minimum of 3 phantom limb pain episodes each week in one phantom leg.
* Degree of pain evaluated by VAS scoring a minimum of 3 cm at time of screening for entry into study.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* Age less than 18 or greater than 70.
* Unilateral upper or lower limb amputation.
* Severe traumatic brain injury (TBI) - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening which is currently performed routinely on patients by the TBI program at WRAMC and noted in the patient's medical record. Subjects with diagnosis of mild TBI following TBI testing, but with a normal score (>42) on the Test of Memory Malingering (TOMM) (parts 1 or 2) can be included in the study.
* Known uncontrolled systemic disease- known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Concurrent participation in another investigational drug or device study for phantom limb pain or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Significant Axis I or II diagnosis determined by a neurologist in the 6 months prior to entry into the study, defined as a condition requiring initiation of medications or hospitalization with continuing medical treatment for the condition.
* Subjects with lack of effort as determined by the neurologist. Subjects will be screened for effort using the TOMM first in order to exclude those with blatant exaggeration or malingering.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Significant decrease in the level of phantom limb pain at 4 weeks. | 4 weeks

SECONDARY OUTCOMES:
Significant decrease in the number and duration of daily phantom limb pain episodes at 4 weeks. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack W Tsao, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Carlen PL, Wall PD, Nadvorna H, Steinbach T. Phantom limbs and related phenomena in recent traumatic amputations. Neurology. 1978 Mar;28(3):211-7. doi: 10.1212/wnl.28.3.211. PMID 564474
- [Background] Manchikanti L, Singh V. Managing phantom pain. Pain Physician. 2004 Jul;7(3):365-75. PMID 16858476
- [Background] Katz J, Melzack R. Pain 'memories' in phantom limbs: review and clinical observations. Pain. 1990 Dec;43(3):319-336. doi: 10.1016/0304-3959(90)90029-D. PMID 2293143
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285
- [Background] Cohen LG, Bandinelli S, Findley TW, Hallett M. Motor reorganization after upper limb amputation in man. A study with focal magnetic stimulation. Brain. 1991 Feb;114 ( Pt 1B):615-27. doi: 10.1093/brain/114.1.615. PMID 2004259
- [Background] Elbert T, Flor H, Birbaumer N, Knecht S, Hampson S, Larbig W, Taub E. Extensive reorganization of the somatosensory cortex in adult humans after nervous system injury. Neuroreport. 1994 Dec 20;5(18):2593-7. doi: 10.1097/00001756-199412000-00047. PMID 7696611
- [Background] Kew JJ, Ridding MC, Rothwell JC, Passingham RE, Leigh PN, Sooriakumaran S, Frackowiak RS, Brooks DJ. Reorganization of cortical blood flow and transcranial magnetic stimulation maps in human subjects after upper limb amputation. J Neurophysiol. 1994 Nov;72(5):2517-24. doi: 10.1152/jn.1994.72.5.2517. PMID 7884476
- [Background] Lotze M, Grodd W, Birbaumer N, Erb M, Huse E, Flor H. Does use of a myoelectric prosthesis prevent cortical reorganization and phantom limb pain? Nat Neurosci. 1999 Jun;2(6):501-2. doi: 10.1038/9145. No abstract available. PMID 10448212
- [Background] Lotze M, Montoya P, Erb M, Hulsmann E, Flor H, Klose U, Birbaumer N, Grodd W. Activation of cortical and cerebellar motor areas during executed and imagined hand movements: an fMRI study. J Cogn Neurosci. 1999 Sep;11(5):491-501. doi: 10.1162/089892999563553. PMID 10511638
- [Background] Birbaumer N, Lutzenberger W, Montoya P, Larbig W, Unertl K, Topfner S, Grodd W, Taub E, Flor H. Effects of regional anesthesia on phantom limb pain are mirrored in changes in cortical reorganization. J Neurosci. 1997 Jul 15;17(14):5503-8. doi: 10.1523/JNEUROSCI.17-14-05503.1997. PMID 9204932
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] Grusser SM, Winter C, Muhlnickel W, Denke C, Karl A, Villringer K, Flor H. The relationship of perceptual phenomena and cortical reorganization in upper extremity amputees. Neuroscience. 2001;102(2):263-72. doi: 10.1016/s0306-4522(00)00491-7. PMID 11166112
- [Background] Ramachandran VS, Rogers-Ramachandran D, Stewart M. Perceptual correlates of massive cortical reorganization. Science. 1992 Nov 13;258(5085):1159-60. doi: 10.1126/science.1439826. No abstract available.
- [Background] Lotze M, Flor H, Grodd W, Larbig W, Birbaumer N. Phantom movements and pain. An fMRI study in upper limb amputees. Brain. 2001 Nov;124(Pt 11):2268-77. doi: 10.1093/brain/124.11.2268. PMID 11673327
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Franz EA, Ramachandran VS. Bimanual coupling in amputees with phantom limbs. Nat Neurosci. 1998 Oct;1(6):443-4. doi: 10.1038/2161. No abstract available. PMID 10196540
- [Background] Jackson PL, Lafleur MF, Malouin F, Richards CL, Doyon J. Functional cerebral reorganization following motor sequence learning through mental practice with motor imagery. Neuroimage. 2003 Oct;20(2):1171-80. doi: 10.1016/S1053-8119(03)00369-0. PMID 14568486
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Bone M, Critchley P, Buggy DJ. Gabapentin in postamputation phantom limb pain: a randomized, double-blind, placebo-controlled, cross-over study. Reg Anesth Pain Med. 2002 Sep-Oct;27(5):481-6. doi: 10.1053/rapm.2002.35169. PMID 12373695